CLINICAL TRIAL: NCT05123196
Title: A Randomized, Double-Blind, Placebo-Controlled, Exploratory Study of MT-8554 in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: Exploratory Study of MT-8554 in Subjects With Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-8554-A-201; jRCT2051210097 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2021-10-18; First posted 2021-11-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Painful Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT-8554 (Experimental): MT-8554 will be started from a low dose, and gradually increase the dose in order.
  Interventions: Drug: MT-8554
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-8554 — Oral Capsule
  Other Names: Elismetrep
  Arms: MT-8554
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, tolerability and pharmacokinetics of MT-8554, compared to placebo, in subjects with painful diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with written consent
2. Patients aged >=20 years at the time of consent
3. Outpatients
4. Patients with pain associated with peripheral symmetric polyneuropathy due to diabetes mellitus and pain lasting >=3 months on the first day of the run-in period. The patient should meet >=2 of the following criteria or nerve conduction studies showing abnormalities in at least one test item (Conduction velocity, amplitude, and latency) for at least two nerves by the first day of run-in period.

   * 1. Subjective symptoms* thought to be due to diabetic polyneuropathy
   * 2. Decreased or eliminated bilateral Achilles tendon reflexes
   * 3. Bilateral decreased vibratory sense of the medial malleolus (=< 10 seconds with a C 128 tuning fork)

     *Subjective symptoms thought to be due to diabetic neuropathy meet the following 3 criteria.
   * Bilateral
   * Toe and plantar symptoms (Numbness, pain or dysesthesia)
   * Does not cause upper extremity symptoms alone
5. Patients whose NRS during the run-in period is assessed for >=4 days of the 7 days immediately before the first day of the treatment period and whose baseline 24-hour mean NRS score is >=4 and =<8.
6. Patients whose rate of change in the 24-hour mean NRS score during the 7 days immediately before the first day of the treatment period is <30%.
7. Patients whose treatment for diabetes mellitus is consistent >=8 weeks before the run-in period, who can consistently maintain the treatment throughout the study period, and in whom the investigator (or sub-investigator) can determine that glycemic control is constant.

Exclusion Criteria:

1. Patients with pain, disease, or skin condition that, in the opinion of the investigator (or sub-investigator), would influence the evaluation of painful diabetic peripheral neuropathy.

   For example, if other pain is in the same location as painful diabetic peripheral neuropathy, or if the pain intensity of the other pain is greater than that of painful diabetic peripheral neuropathy, which in the opinion of the investigator (or sub-investigator) would impact the assessment of painful diabetic peripheral neuropathy.
2. Patients who have had amputation of upper and lower limbs other than toes due to gangrene caused by impaired blood circulation.
3. Patients who do not meet the criteria of prohibited concomitant drugs or restricted concomitant drugs.
4. Patients with hypersensitivity to acetaminophen or a history of hypersensitivity to acetaminophen.
5. Patients with New York Heart Association functional class III or IV symptoms of heart failure.
6. History of myocardial infarction, congestive heart failure, unstable angina, or cerebrovascular disorder (excluding lacunar infarction) within 6 months prior to informed consent.
7. Patients with major psychiatric disorder such as depression or anxiety disorder.
8. Patients with drug abuse or a history of drug abuse.
9. Patients with current or previous infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). However, patients with previous infection with hepatitis B virus who are HBsAg-negative are eligible.
10. Patients with HbA1c > 10.5%.
11. Patients with poorly controlled hypertension (>= 180 mmHg systolic and/or >= 110 mmHg diastolic).
12. Patients with eGFR < 30 mL/min/1.73 m^2.
13. Patients with AST or ALT > 2.5*ULN.
14. Patients who answered "Yes " to any item of Columbia Suicide Severity Rating Scale within the past 12 months.
15. Patients who have a concomitant malignancy or a history of malignancy. However, patients who have a history of malignancy but have not experienced recurrence for at least 5 years before informed consent (patients who have not experienced recurrence for at least 5 years after the last administration if the patients were receiving anticancer drugs) will be excluded.
16. Male or female patients of childbearing potential who do not agree to use contraception from the date of informed consent until 3 months after the completion (discontinuation) of investigational product.
17. Female patients who are pregnant, breastfeeding or possibly pregnant.
18. Patients who participated in another clinical study and received investigational product within 12 weeks before informed consent.
19. Prior exposure to MT-8554.
20. Other patients who, in the opinion of the investigator (or sub-investigator), are ineligible for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the weekly mean 24-hour average NRS score at Week 12 in treatment period | Baseline and Week 12
  Numeric Rating Scale (NRS) is the 11-point numerical rating scale of 0 (no pain) to 10 (worst possible pain). Higher NRS scores indicated worse outcome.

SECONDARY OUTCOMES:
Change from baseline in weekly mean 24-hour average NRS score at each assessment point | Up to Week 12
  Numeric Rating Scale (NRS) is the 11-point numerical rating scale of 0 (no pain) to 10 (worst possible pain). Higher NRS scores indicated worse outcome.
Average weekly 24-hour NRS score during the 12 week treatment period 30% and 50% responder rates | Baseline and Week 12
  Numeric Rating Scale (NRS) is the 11-point numerical rating scale of 0 (no pain) to 10 (worst possible pain). Higher NRS scores indicated worse outcome.
Change from baseline in weekly mean daily NRS score at each assessment point | Up to Week 12
  Numeric Rating Scale (NRS) is the 11-point numerical rating scale of 0 (no pain) to 10 (worst possible pain). Higher NRS scores indicated worse outcome.
Change from baseline in weekly mean nocturnal average NRS score at each assessment point | Up to Week 12
  Numeric Rating Scale (NRS) is the 11-point numerical rating scale of 0 (no pain) to 10 (worst possible pain). Higher NRS scores indicated worse outcome.
Change from baseline in weekly mean 24 hour worst NRS score at each assessment point | Up to Week 12
  Numeric Rating Scale (NRS) is the 11-point numerical rating scale of 0 (no pain) to 10 (worst possible pain). Higher NRS scores indicated worse outcome.
Change from baseline in NPSI at each assessment point | Up to Week 12
  Neuropathic Pain Symptom Inventory (NPSI) is the questionnaire to evaluate the different symptoms of neuropathic pain and each symptoms are evaluated from 0 (no pain) to 10 (worst possible pain). Higher NPSI scores indicated worse outcome.
Change from baseline in BPI pain severity at each assessment point | Up to Week 12
  Brief Pain Inventory (BPI) is the questionnaire to assess the severity of pain from 0 (no pain) to 10 (pain as bad as patient can imagine). Higher BPI scores indicated worse outcome.
Change from baseline in BPI functional impairment at each assessment point | Up to Week 12
  Brief Pain Inventory (BPI) is the questionnaire to assess the impact of pain on daily functions from 0 (does not interfere) to 10 (completely interferes). Higher BPI scores indicated worse outcome.
Change from baseline in MOS-SS at each assessment point | Up to Week 12
  Medical Outcomes Study-Sleep Scale (MOS-SS) is the questionnaire to evaluate the "sleep disorder " "snoring" "sleep arousal with shortness of breath or headache" "sleep sufficiency" "somnolence" and "amount of sleep/optimal sleep" ranges from 0 (all of the time) to 6 (none of the time). Lower MOS-SS scores indicated worse outcome.
Proportion of PGIC responders at each assessment point | Up to Week 12
  Patient Global Impression of Change (PGIC) is a questionnaire to evaluate the overall impression of pain improvement by patient from 1 (very much improved) to 7 (very much worse). Higher PGIC scores indicated worse outcome.
Proportion of CGIC responder at each assessment point | Up to Week 12
  Clinician Global Impression of Change (CGIC) a questionnaire to evaluate the overall impression of pain improvement by clinician from 1 (very much improved) to 7 (very much worse). Higher CGIC scores indicated worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (33):
- Japan (33):
  - Yachiyo Hospital, Anjo, Aichi-ken
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital, Nagoya, Aichi-ken
  - JUNEIKAI Medical Corporation Akaicho Clinic, Chiba, Chiba
  - Social Medical Corporation the Chiyukai foundation Fukuoka Wajiro Hospital, Fukuoka, Fukuoka
  - TOJITAMA thyroid and diabetes Clinic, Fukuoka, Fukuoka
  - Kunisaki Makoto Clinic, Fukuoka, Fukuoka
  - Steel Memorial Yawata Hospital, Kitakyushu-shi, Fukuoka
  - Medical Corporation Kouhoukai Takagi Hospital, Okawa-shi, Fukuoka
  - Matsunami Health Promotion Clinic, Hashima-gun, Gifu
  - Kikuchi Clinic of Internal Medicine, Maebashi, Gunma
  - Japanese Red Cross Asahikawa Hospital, Asahikawa, Hokkaido
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Jiyugaoka Yamada Internal Medicine Clinic, Obihiro, Hokkaido
  - Sanuki Municipal Hospital, Sanuki-shi, Kagawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa-shi, Kanagawa
  - Shunkaikai Inoue Hospital, Nagasaki, Nagasaki
  - Medical Corporation Keiaikai Nakamura Hospital, Beppu, Oita Prefecture
  - Medical Corporation Ikeikai Inobe Funai Clinic, Ōita, Oita Prefecture
  - Abe Diabetes Clinic, Ōita, Oita Prefecture
  - Saiki Central Hospital, Saiki, Oita Prefecture
  - Medical Corporation Heishinkai OCROM Clinic, Suita, Osaka
  - Hisatomi Clinic, Saga, Saga-ken
  - Soka Sugiura Internal Medicine Clinic, Sōka, Saitama
  - OMI MEDICAL CENTER, Social Medical Corporation Seikoukai, Kusatsu, Shiga
  - Kumanomae Nishimura Naika Clinic, Arakawa-ku, Tokyo
  - Tokyo Center Clinic, Chuo-ku, Tokyo
  - Sugawara Clinic, Nerima-ku, Tokyo
  - Ome Municipal General Hospital, Ome-shi, Tokyo
  - Medical Corporation Souaikai Aihara Medical Clinic, Shinagawa-ku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku, Tokyo
  - Japan Organization of Occupational Health and Safety Sanin Rosai Hospital, Yonago, Tottori
  - Kitano Hospital, Tazuke Kofukai Medical Research Institute, Osaka

IPD SHARING:
Plan to Share IPD: Yes
When requested by a qualified researcher in the field of science or medicine, Tanabe Pharma Corporation will share clinical trial data that was collected from individual patients in a clinical trial with that researcher after a review committee of experts determines that such sharing is appropriate.
  Access Criteria: Please refer to the following link for conditions and limitations for sharing data.
  URL: https://www.tanabe-pharma.com/en/develop/protocol.html